CLINICAL TRIAL: NCT04617847
Title: A Multicenter, Open-label Extension Study to Evaluate the Safety, Pharmacodynamics, and Clinical Effects of WVE-120101 in Patients With Huntington's Disease
Brief Title: Open-label Extension Study to Evaluate the Safety and Tolerability of WVE-120101 in Patients With Huntington's Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVE-HDSNP1-002
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- WVE-120101 (Dose A) (Experimental)
  Interventions: Drug: WVE-120101

INTERVENTIONS:
Drug: WVE-120101 — WVE-120101 is a stereopure antisense oligonucleotide (ASO). It is administered monthly via intrathecal injection.

SUMMARY:
WVE-HDSNP1-002 is an open-label extension (OLE) study to evaluate the safety, tolerability, PK, PD, and clinical effects of WVE-120101 in adult patients with early manifest HD who carry a targeted single nucleotide polymorphism, rs362307 (SNP1). To participate in the study, patients must have completed the Phase 1b/2a clinical study WVE-HDSNP1-001.

ELIGIBILITY:
Key Inclusion Criteria:

* 1. Patient successfully completed the Phase 1b/2a study with WVE-120101, WVE-HDSNP1-001.

Key Exclusion Criteria:

* 1. Received an investigational drug other than WVE-120101, including an investigational oligonucleotide, within the past 1 year or 5 half-lives of the drug, whichever is longer.
* 2. Inability to undergo brain MRI (with or without sedation).
* 3. Clinically significant medical finding on the physical examination other than HD that, in the judgment of the Investigator, will make the patient unsuitable for participation in and/or completion of the study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Wave Life Sciences
Locations (18):
- Australia (7):
  - Westmead Hospital, Sydney, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Royal Melbourne Hospital, Carlton, Victoria
  - Monash Health, Clayton, Victoria
  - Alfred Health, Melbourne, Victoria
  - Calvary Health Care Bethlehem, Parkdale, Victoria
  - North Metropolitan Health Service, Perth, Western Australia
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Centre Hospitalier de l-Universite de Montreal, Montreal, Quebec
- Denmark (2):
  - Aarhus Universitets Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (2):
  - Hospital Henri Mondor, Créteil
  - Institut du Cerveau et de la Moelle Epinière, Paris
- George-Huntington-Institut GmbH, Münster, Germany
- Poland (2):
  - Szpital Sw. Wojciecha, Gdansk
  - Instytut Psychiatrii i Neurologii, Warsaw
- United Kingdom (2):
  - Royal Devon and Exeter Hospital NHS Trust, Exeter, Devon
  - Queen Elizabeth University Hospital - PPDS, Glasgow, Glasgow City

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the original OLE study protocol, patients who were in the 2 and 4 mg dose cohorts in the Phase 1b/2a study were to be enrolled into the 4 or 8 mg dose group in this study. Patients in the 8 and 16 mg dose cohorts in WVE-HDSNP1-001 continued to receive that dose. As of Amendment 1.0 of this protocol, all new patients were to be enrolled at a dose level of at least 16 mg. All current patents were dose modified to 16 or 32 mg.
Groups:
- 4 mg WVE-120101: Enrolled at 4 mg WVE-120101 dose level
- 16 mg WVE-120101: Enrolled at 16 mg WVE-120101 dose level
Period: Overall Study
Arm/Group | 4 mg WVE-120101 | 16 mg WVE-120101
Started | 3 | 24
Dose Modified to 16 mg WVE-120101 | 3 | 1
Dose Modified to 32 mg WVE-120101 | 0 | 5
Completed | 0 | 0
Not Completed | 3 | 24
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 2
Not completed — Death | 0 | 1
Not completed — Termination of Study by Sponsor | 2 | 21

BASELINE CHARACTERISTICS:
Groups:
- 16 mg WVE-120101: Enrolled at 12 mg WVE-120101 dose level
- Total: Total of all reporting groups
Arm/Group | 4 mg WVE-120101 | 16 mg WVE-120101 | Total
Number analyzed (Participants) | 3 | 24 | 27
Age, Categorical [Count of Participants; unit: Participants] — Demographics at the time of enrollment in the WVE-HDSNP1-001 study.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 3 | 24 | 27
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 15 | 17
  Male | 1 | 9 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 24 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 24 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 3 | 6
  Denmark | 0 | 2 | 2
  Poland | 0 | 9 | 9
  Australia | 0 | 8 | 8
  France | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Patients With Treatment-emergent AEs (TEAEs)
Time Frame: First dose received (Day 1) through the Study Termination visit (maximum of 45 weeks of treatment)
Population: Patients treated at more than one dose level (e.g., initial dose and after dose modification) are included in each applicable dose group. Adverse events are counted in the dose the patient was receiving at the time of onset.
Measure: Count of Participants; unit: Participants
Groups:
- 4 mg WVE-120101: Patients who received 4 mg WVE-120101 at any point in the study
- 16 mg WVE-120101: Patients who received 16 mg WVE-120101 at any point in the study
- 32 mg WVE-120101: Patients who received 32 mg WVE-120101 at any point in the study
Arm/Group | 4 mg WVE-120101 | 16 mg WVE-120101 | 32 mg WVE-120101
Number analyzed (Participants) | 3 | 27 | 5
Participants | 2 | 17 | 2

2. Primary Outcome: Safety: Number of Patients With a Severe TEAE
Time Frame: First dose received (Day 1) through the Study Termination visit (maximum of 45 weeks of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg WVE-120101 | 16 mg WVE-120101 | 32 mg WVE-120101
Number analyzed (Participants) | 3 | 27 | 5
Participants | 0 | 5 | 0

3. Primary Outcome: Safety: Number of Patients With Serious TEAEs
Time Frame: First dose received (Day 1) through the Study Termination visit (maximum of 45 weeks of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg WVE-120101 | 16 mg WVE-120101 | 32 mg WVE-120101
Number analyzed (Participants) | 3 | 27 | 5
Participants | 0 | 3 | 1

4. Primary Outcome: Safety and Tolerability: Number of Patients Who Withdraw Due to TEAEs
Time Frame: First dose received (Day 1) through the Study Termination visit (maximum of 45 weeks of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg WVE-120101 | 16 mg WVE-120101 | 32 mg WVE-120101
Number analyzed (Participants) | 3 | 27 | 5
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: First dose received (Day 1) through the Study Termination visit (maximum of 45 weeks of treatment)
Arm/Group | 4 mg WVE-120101 | 16 mg WVE-120101 | 32 mg WVE-120101
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/27 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/27 | 1/5
Other Adverse Events (participants affected / at risk) | 2/3 | 16/27 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 mg WVE-120101 (N=3) | 16 mg WVE-120101 (N=27) | 32 mg WVE-120101 (N=5)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Completed Suicide (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 4 mg WVE-120101 (N=3) | 16 mg WVE-120101 (N=27) | 32 mg WVE-120101 (N=5)
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 3 | 0
CSF Protein Increased (Investigations) | 1 | 1 | 0
CSF white blood cell count increased (Investigations) | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 7 | 0
Headache (Nervous system disorders) | 0 | 5 | 0
Dysarthria (Nervous system disorders) | 0 | 2 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/47/NCT04617847/Prot_SAP_000.pdf